CLINICAL TRIAL: NCT03310515
Title: A Cohort Study to Determine the Incidence of HIV-1 Infection in HIV-1 Uninfected High Risk Participants Who Are Male Sex at Birth and Have Sex With Men
Brief Title: Incidence of Human Immunodeficiency Virus-1 (HIV-1) Infection in HIV-1 Uninfected High Risk Men Who Have Sex With Men
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 206897
Record Dates: First submitted 2017-09-21; First posted 2017-10-16 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: PrEP; MSM; seroincidence; HIV-1; TGW; STIs
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-1 uninfected high risk subjects: The study will involve HIV-1 uninfected high risk MSM and TGW subjects. They will receive comprehensive prevention package including HIV and safe sex counseling, provision of condoms and water-based lubricant, and STI screening and referral for treatment. Visits will include Baseline screening for HIV followed by screenings at Day 1, Weeks 5, 9, and 8 week intervals thereafter until study conclusion. Screening for other STIs will occur at Baseline, Week 9, and every 16 weeks thereafter.
  Interventions: Behavioral: Risk reduction counseling; Other: Social harm interview; Other: Computer-Assisted Self Interviewing technique

INTERVENTIONS:
Behavioral: Risk reduction counseling — Subjects will receive comprehensive prevention package including HIV and safe sex counseling, provision of condoms and water-based lubricant, and STI screening and referral for treatment.
Other: Social harm interview — Information regarding social harms (loss of privacy, stigmatization, interference with gainful employment, and coercion) will be solicited during bi-monthly study visits after enrollment in the study and will be recorded. Subjects who report social harms will be referred to speak with a social worker and/or a study counselor.
Other: Computer-Assisted Self Interviewing technique — Demographic, behavioral, and psychosocial factors associated with HIV acquisition will be assessed by CASI.

SUMMARY:
Studies to assess the effectiveness of interventions to prevent HIV infection depend upon robust estimates of Baseline HIV incidence rates. The changing landscape of high-risk populations, as well as the evolution of biomedical pre-exposure prophylaxis (PrEP) interventions, requires a contemporary evaluation of HIV incidence as well as demographic, behavioral and other subject factors which may impact HIV incidence. This is a prospective cohort study to measure HIV-1 seroincidence in a study population of HIV-1 uninfected Chinese men who have sex with men (MSM) and transgender women (TGW) who are at high-risk of HIV infection. Approximately 550 subjects who are male sex at birth and have sex with men shall enter the study, which will allow for a 10% drop out rate to maintain 500 subjects at the conclusion of the cohort. This is a single arm cohort study to determine HIV-1 seroincidence rates in high risk MSM and TGW when combined with a comprehensive prevention package including HIV and safe sex counseling, provision of condoms and water-based lubricant, and sexually transmitted infection (STI) screening and referral for treatment. It will be determined what proportion of high-risk MSM and TGW who are given a comprehensive HIV-1 prevention package will acquire HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are Chinese MSM and/or TGW and must be 18 years or older at the time of screening.
* Subjects of male sex at birth and who have sex with men, who in the 6 months prior to screening report one or more of the following risk criteria:

  * Unprotected (condomless) receptive anal intercourse with one or more partners.
  * More than five partners in the 6 months prior to enrolment (regardless of condom use and HIV serostatus, as reported by the enrolee).
  * Reported STI with syphilis, gonorrhea, chlamydia, chancroid, or lymphogranuloma venereum.

Subjects in a monogamous relationship with an HIV-1 seronegative partner or a virologically-suppressed HIV-1 + partner for >1 year are not eligible for participation.

* Males, agree to appropriate use of contraceptive measures during heterosexual intercourse.
* Subjects who have non reactive fourth generation HIV test and undetectable HIV-1 RNA at screening.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Subjects with known moderate to severe hepatic impairment as per liver function test criteria outlined below.
* Subject who, in the investigator's judgment, poses a significant suicide risk.
* The Subject has a tattoo or other dermatological condition overlying the gluteus region.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Use of PrEP or post exposure prophylaxis (PEP) within the last 30 days prior to screening.
* Current use or anticipated need for use high dose aspirin or other anticoagulants including antiplatelet medications that would interfere with the ability to receive intramuscular (IM) injections.
* Exposure to an experimental drug and/or experimental vaccine within 28 days or 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the screening.
* Anti-tuberculosis therapy.
* Alcohol use that in the judgment of the investigator would interfere with the subject's ability to complete study procedures.
* Active injection drug use that in the judgment of the investigator would interfere with the subject's ability to complete study procedures.
* Any medical condition, including psychiatric conditions, that in the judgment of the investigator would interfere with the subject's ability to complete study procedures.
* A reactive HIV test at screening.
* A positive Hepatitis B surface antigen.
* A positive Hepatitis C antibody with an HCV viral ribose nucleic acid (RNA) above the lower limit of detection.
* Any of the following laboratory values at screening:

  * Hemoglobin (Hgb) <11 gram per deciliter (g/dL).
  * Absolute neutrophil count <750 cells per cubic millimeter (cells/mm^3).
  * Platelet count <100,000 cells/mm^3.
  * Presence of a coagulopathy defined by an international normalized ratio (INR)>1.5 or a partial thromboplastin time (PTT)>45 seconds.
  * Creatinine clearance <60 milliliter per minute (mL/min) using the Cockroft-Gault equation.
  * Aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN).
  * Direct Bilirubin >2.0 milligram per deciliter (mg/dL).
* Co-enrolment in any other HIV interventional studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Chinese MSM and/or TGW will be enrolled.
Study Population: This prospective cohort study will involve population of HIV-1 uninfected Chinese MSM and TGW who are at high-risk of HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
HIV-1 seroincidence rate in a cohort of high-risk MSM and TGW | Baseline, Day 1, Weeks 5, 9, and every 8 week intervals thereafter until study completion, an average of 12 months
  Incidence of HIV-1 infection in subject's post-study entry will be assessed by determining number of subjects who become infected with HIV-1 post-screening and after study entry including Day 1 and subsequent observation visits. Confirmatory HIV serology test will be performed at seroconversion visit.
HIV-1 seroincidence rate in a cohort of high-risk TGW | Baseline, Day 1, Weeks 5, 9, and every 8 week intervals thereafter until study completion, an average of 12 months
  Incidence of HIV-1 infection in subject's post-study entry will be assessed by determining number of subjects who become infected with HIV-1 post-screening and after study entry including Day 1 and subsequent observation visits. Confirmatory HIV serology test will be performed at seroconversion visit.

SECONDARY OUTCOMES:
Number of subjects diagnosed with gonorrhea, chlamydia, and syphilis post screening | Day 1, Week 9, and every 16 weeks interval thereafter until study completion, an average of 12 months
  Infections like gonorrhea, chlamydia, and syphilis will be assessed by toluidine red unheated serum test (TRUST) for syphilis and STI testing.
Number of subjects with demographic factors | Day 1, Week 9, and every 8 weeks interval thereafter until study completion, an average of 12 months
  Demographic factors associated with HIV seroconversion and STI acquisition will be assessed by computer-assisted self-interview (CASI).
Number of subjects enrolled and retained in to the study | Day 1, Weeks 5, 9, and every 8 or 16 weeks interval thereafter until study completion, an average of 12 months
  Measures will be utilized to effectively engage and retain the subjects in the study. Retention strategies to be studied may include community engagement, interpersonal relationship building and reduction of external barriers.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (8):
- China (8):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenzhen